CLINICAL TRIAL: NCT02221661
Title: Non-interventional Longitudinal Study in Alzheimer Disease Diagnosis in Primary Consultants Patients With Cognitive and / or Memory Complaint Requiring Specialized Exploration Using AclarusDx® Blood Test in Memory Centers
Brief Title: Performance of AclarusDx® a Blood-Based Transcriptomic Test for AD, in French Patients Newly Referred to a Memory Center
Acronym: DIALOG
Status: Completed | Type: Observational
Sponsor: Diaxonhit (Industry)
Collaborators: Olivier SOL, MD (Unknown)
Responsible Party: Sponsor
Other Study IDs: MG/JD/11.830
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Cognitive Impairment; Memory Complaint; Clinical Investigation in Memory Centers
Keywords: Alzheimer; cognitive impairment; blood test
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Whole blood samples collected in PAXgene® blood RNA tubes
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the performance of AclarusDx™, an investigational blood test detecting gene expression information, and intended to help physicians in making an Alzheimer's Disease diagnosis in patients having memory complaint and/or cognitive impairments.

DETAILED DESCRIPTION:
The objective of this study is to apply AclarusDx™ signature in 600 patients newly referred in french memory centers. Only AclarusDx™ will be added to the panel of tests usually performed at the centers to establish diagnosis. AclarusDx™ will be used for investigational use only, not for diagnostic purpose. The ultimate goal is to define the clinical utility of AclarusDx™ to provide physicians with a tool that will help them in making the diagnosis of Alzheimer's Disease (AD).

The primary objective is to estimate the prevalence of positive AclarusDx™ in patients diagnosed AD in the population of primary consultants. This population of primary consultants consists of patients with cognitive impairment and / or a memory complaint requiring specialized exploration using AclarusDx™ blood test and which may be potentially related to multiple and different etiologies.

The secondary objectives are:

* Assess the prevalence of positive AclarusDx™ in relation to other diagnoses (MCI, vascular dementia ...) established by the physician investigator at the end of specialized assessment.
* Identify the demographic factors anamnestic, clinical, biological and imaging associated with positivity of AclarusDx™
* Identify the demographic factors anamnestic, clinical, biological and imaging associated with the diagnosis of AD and other diagnoses.
* Determine the contribution of AclarusDx™ in the usual battery of tests performed for diagnostic approach to Alzheimer's disease and to identify a possible association of interest with one or more endpoints (clinical, neuropsychological, brain, biological imaging).
* Assess: diagnostic status at 6 and 12 months, and the MMSE and IADL at 6 and 12 months.
* assess the predictive value of AclarusDx™ achieved during the initial visit to the diagnosis of AD is 12 months.
* Evaluate AclarusDx™ predictive value to 12 months

ELIGIBILITY:
Inclusion Criteria:

* male and female adult patients
* suffering from cognitive impairment and/or memory complaint and justifying a first clinical investigation at the memory center

Exclusion Criteria:

* patient already followed up by the memory center
* patient unable to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cognitive impairment and/or memory complaint justifying a first clinical investigation for diagnosis
Sampling Method: Probability Sample
Enrollment: 606 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Estimation of the prevalence of positive AclarusDx™ among patients clinically AD diagnosed | Outcome measured during one single study visit
  The primary outcome is to estimate the prevalence of positive AclarusDx Alzheimer patients diagnosed (excluding MCI).
  The prevalence is estimated as a percentage calculated among patients being confirmed clinically as having AD at the Memory Center and having a positive or negative AclarusDx™ result